CLINICAL TRIAL: NCT03816293
Title: SUpPress SSI - Single Use Negative Pressure Wound Therapy (NPWT) to Reduce Surgical Site Infections
Acronym: SUpPressSSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Iowa (Other); University of Maryland (Other); Emory University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); Acelity (Other)
Responsible Party: Principal Investigator, Susan Casey Bleasdale, Associate Professor of Clinical Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2018-1300; U01CK000557-01-00 (Other Grant/Funding Number: CDC); U01CK000557-01 (NIH)
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Surgical Site Infection; Obesity; Diabetes; Cesarean Section Complications
Keywords: colon surgery; abdominal hysterectomy
MeSH Terms: conditions — Surgical Wound Infection; Obesity; Diabetes Mellitus | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Randomized stepped wedge cluster but site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Negative Pressure Wound Therapy (Active Comparator): NPWT use on closed incision for 7 days after c-section, abdominal hysterectomy, and colon surgery in patients with diabetes and/or obesity
  Interventions: Device: Negative Pressure Wound Therapy
- Control Dressing (No Intervention): Standard dressing on closed incisions after c-section, abdominal hysterectomy, and colon surgery in patients with diabetes and/or obesity

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — Occlusive dressing with attached Prevena incision management with 125mmHg of negative pressure and cartridge to manage secretions
  Other Names: Prevena Incision Management
  Arms: Negative Pressure Wound Therapy

SUMMARY:
Our goal is to provide data that will give surgeons and hospitals clear recommendations on the use of NPWT for Cesarean section, abdominal hysterectomy and colon surgeries in patients with diabetes and/or obesity. We also want to understand the patient experience with the dressing so that we can provide information that will enable clinicians to remove barriers to NPWT use. Additionally, we are seeking to use automated electronic medical record decision support to identify patients that will benefit most from the NPWT.

DETAILED DESCRIPTION:
Specific Aim 1: Evaluate the effect of single-use NPWT on SSI rates after C-section, abdominal hysterectomy, and colon procedures in at risk patients.

To address this aim, we will conduct multicenter, stepped-wedge, quasi-experimental trial evaluating use of the PrevenaTM with 125 mm Hg negative pressure for 7 days among obese (BMI >30) and/or diabetic patients undergoing the procedures of interest. This is essentially a phase IV clinical trial as this dressing has FDA approval for the indicated use.

Specific Aim 2: Investigate the patients' experience of using the NPWT. To achieve this aim, we will survey a sub-set of patients to assess their knowledge of post-operative care, to identify complications associated with NPWT use, and to learn how patients evaluated the device's ease of use, ease of removal, and comfort.

Specific Aim 3: Assess whether real-time decision support through machine-learning modeling can help surgeons identify patients at high risk of SSI who could benefit from NWPT or other post-surgical preventive measures. To address this aim, we will evaluate whether boosted tree modeling techniques can be used "at the bedside" via electronic medical record data feeds to tailor post-operative care and preventive care for specific patients.

ELIGIBILITY:
Inclusion Criteria: Category A and B

A. Patients undergoing any of the below procedures:

1. C-section
2. abdominal hysterectomy
3. colon procedures Surgical procedures selected will be based on NHSN designated ICD-10 PCS codes(14), with the exclusion of laparoscopic procedures.

B. and either of the following medical conditions:

1. obesity, BMI >30 kg/m2
2. diabetes type 1 or 2 Criteria for a diagnosis of diabetes: Diabetes noted in the problem list or the medical history or Patient is taking a medication as treatment for diabetes, consistent with NHSN criteria(10).

Exclusion Criteria:

1. Age less than 18 years
2. Infection present at the time of the surgery
3. Laparoscopic procedures with incisions <6cm.
4. Patients using alternative NPWT device other than the PrevenaTM with 125 mm Hg negative pressure
5. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3680 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection Rate per 100 surgeries | within 30 days after surgery
  Superficial , Deep and organ space infections after surgery

SECONDARY OUTCOMES:
Post Operative Length of Stay (days) | within 30days after surgery
  days of ongoing admission after surgery
REadmission incidence and rate per 100 surgeries | within 30 days
  REadmission to hospital after discharge from surgery
Seroma incidence and rate per 100 surgeries | with in 30 days after surgery
  Non infectious Fluid accumulation
Hematoma incidence and rate per 100 surgeries | within 30 days after surgery
  Bloody fluid collection
Dehiscence incidence and rate per 100 surgeries | within 30 days after surgery
  Loss of incision apposition

CONTACTS AND LOCATIONS:
Overall Officials: Susan Bleasdale, MD, Principal Investigator — University of Illinois at Chicago
Locations (5):
- United States (5):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - University of Illinois Hospital, Chicago, Illinois
  - University of Iowa Health System, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
This is a study with waiver of consent data will be in aggregate without patient identifiers